CLINICAL TRIAL: NCT03527875
Title: Process Optimization of Preoperative Biliary Drainage in Patients With Malignant Obstructive Jaundice of Extrahepatic Bile Duct: A Multi-center, Prospective, Open-labeled, Real World Study Based on Electronic Data Capture System
Brief Title: Process Optimization of Preoperative Biliary Drainage in Patients With Malignant Obstructive Jaundice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018ZSLC24
Record Dates: First submitted 2018-04-23; First posted 2018-05-17 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Jaundice, Obstructive; Klatskin Tumor
MeSH Terms: conditions — Jaundice, Obstructive; Klatskin Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PTBD group (Experimental): Percutaneous Transhepatic Biliary Drainage
  Interventions: Procedure: PTBD group
- ENBD group (Experimental): Endoscopic Nasobiliary Biliary Drainage
  Interventions: Procedure: ENBD group
- EBS group (Experimental): Endoscopic Biliary Stenting
  Interventions: Procedure: EBS group
- Without PBD group (No Intervention): receive surgery without PBD

INTERVENTIONS:
Procedure: PTBD group — Percutaneous Transhepatic Biliary Drainage, a kind of Preoperative Biliary Drainage methods for hilar cholangiocarcinoma patients
  Arms: PTBD group
Procedure: ENBD group — Endoscopic Nasobiliary Drainage, a kind of Preoperative Biliary Drainage methods for hilar cholangiocarcinoma patients
  Arms: ENBD group
Procedure: EBS group — Endoscopic Biliary Stenting, a kind of Preoperative Biliary Drainage methods for hilar cholangiocarcinoma patients
  Arms: EBS group

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of different methods of preoperative biliary drainage in patients with extrahepatic bile duct neoplasms with obstructive jaundice (hilar cholangiocarcinoma, distal bile duct cancer, and periampullary carcinoma), including PTBD (Percutaneous Transhepatic Biliary Drainage), ENBD (Endoscopic Nasobiliary Drainage) and EBS (Endoscopic Biliary Stenting).

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the following four criteria are included into the study:

  1. Preoperative clinical diagnosis of hilar cholangiocarcinoma, distal bile duct cancer, periampullary cancer without distant metastasis or peripheral vascular invasion, and plan for radical surgery;
  2. Serum total bilirubin is higher than 51 umol/l;
  3. Age is older than 18 and younger than 80 years old;
  4. Sign in informed consent to receive preoperative PTBD, ENBD, EBS or without PBD.

Exclusion Criteria:

* If any of the following items are met, the subject cannot enter the study.

  1. Incorporate severe mental illness, severe heart, lungs and kidneys disease, etc., and be unable to tolerate surgery;
  2. Malignant obstructive jaundice caused by metastatic tumors;
  3. Pregnancy or lactation women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Complication rate after drainage | From PBD to completion of radical surgery, an average of 1 month
  Complication rate between PBD (preoperative biliary drainage) and radical surgery
Complication rate after radical surgery | 1 month post operatively
  Complication rate after radical surgery
Success rate of PBD | Day 1
  Success rate of different methods of PBD

SECONDARY OUTCOMES:
operative time | Day 1
  duration of radical surgery
Hepatoduodenal edema | at time of radical surgery
  Degree of hepatoduodenal edema (including no edema, mild edema, moderate edema, and severe edema)
Perioperative mortality | from PBD to 4 weeks after surgery, an average of 2 month
  Mortality between PBD and 4 weeks after surgery
implantation metastasis | Day 1
  Rate of implantation metastasis
Rate of change in Total bilirubin | 2 weeks after PBD
  Recovery efficiency of liver function
Rate of change in alanine aminotransferase | 2 weeks after PBD
  Recovery efficiency of liver function
Rate of change in aspartate aminotransferase | 2 weeks after PBD
  Recovery efficiency of liver function

IPD SHARING:
Plan to Share IPD: No